CLINICAL TRIAL: NCT02363829
Title: A Phase I Study of Nelfinavir Added to Cisplatin Chemotherapy Concurrent With Pelvic Radiation for Locally Advanced Cervical Cancer (II-IVA)
Brief Title: A Study of Nelfinavir Added to Cisplatin Chemotherapy Concurrent With Pelvic Radiation for Locally Advanced Cervical Cancer (II-IVA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 32814
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Uterine Cervix Cancer
Keywords: clinical stages IIA, IIB, IIIA, IIIB, IVA; invasive carcinoma; uterine cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acidemia, isovaleric | interventions — Nelfinavir; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Nelfinavir and Cisplatin
  Interventions: Drug: Nelfinavir; Biological: Cisplatin

INTERVENTIONS:
Drug: Nelfinavir
Biological: Cisplatin

SUMMARY:
Patients 18 years of age and older with clinical stages IIA, IIB, IIIA, IIIB, IVA cervical carcinoma limited to the pelvis will receive twice daily oral nelfinavir (NFV) and weekly IV cisplatin in combination as radiosensitizers with daily whole pelvic external beam and intracavitary radiation brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary, previously untreated, histologically confirmed invasive carcinoma of the uterine cervix (any cell type). Clinical stages IIA, IIB, IIIA, IIIB, IVA. A representative H & E stained slide showing documentation of the primary invasive cancer is required.
* Patients must have adequate bone marrow, renal and hepatic function:

Laboratory work must be performed within 30 days prior to start of study treatment.

ANC ≥ 1,500/μL; Platelet count ≥ 100,000/μL; Creatinine < 2.0 mg/dL; Total Bilirubin ≤ 1.5 times normal; SGOT ≤ 3 times normal.

* Patients with a ECOG/GOG Performance Status of 0, 1, or 2.
* Patients with ureteral obstruction must be treated with stent or nephrostomy tube.
* Patients of childbearing potential must use an effective form of birth control."Patients receiving oral contraceptives should be instructed that alternate or additional contraceptive measures should be used during therapy with VIRACEPT. "
* Confirmed seronegative HIV status within 3 months prior to start of study treatment.
* Patients must be at least 18 years of age.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.

Exclusion criteria

* Patients with Stage IA, IB or IVB disease.
* Patients who have known metastases to other organs outside the radiation field at the time of the original clinical and surgical staging.
* Patients who have received previous pelvic or abdominal radiation, cytotoxic chemotherapy, or previous therapy of any kind for this malignancy.
* Patients with septicemia or severe infection.
* Patients who have circumstances that will not permit completion of this study or the required follow-up.
* Patients who are pregnant at the time of diagnosis and do not wish pregnancy termination prior to initiation of treatment.
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields.
* Patients with other concomitant malignancies (with the exception of non-melanoma skin cancer), who had (or have) any evidence of other cancer present within the last 5 years.
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Patients with poorly controlled diabetes mellitus despite medication.
* Patients taking anti-arythmic agents such as amiodarone, quinidine, rifampin, ergot derivatives such as ergotamine, St John's Wort, HMG-CoA reductase inhibitors such as lovastatin, neuroleptic such as pimozide, sedatives such as midazolam and triazolam among other CYP3A4 and CYP2C19 substrates.
* Patients with Phenylketonuria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Simpkins, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Lilie Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States